CLINICAL TRIAL: NCT03337841
Title: Neoadjuvant Treatment in the Prevention of Recurrence of Hepatocellular Carcinoma With Pembrolizumab Trial (AURORA)
Brief Title: Pembrolizumab as Neoadjuvant Treatment in HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kindai University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Masatoshi Kudo, Professor, Kindai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AURORA study
Record Dates: First submitted 2017-10-30; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Neo adjuvant chemotherapy; Adjuvant chemotherapy; Immune checkpoint inhibitor; Pembrolizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg IV once only in the neoadjuvant phase. Pembrolizumab 200 mg IV every 3 weeks in the adjuvant phase.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Each subject will receive administration of pembrolizumab 200mg IV once only before curative treatment such as hepatic resection or radiofrequency ablation, and will receive curative treatment after administration of pembrolizumab. After curative treatment, each subject will receive pembrolizumab 200mg IV every 3 weeks. Treatment will continue until tumor recurrence, occurrence of an unacceptable adverse event, or the 16th treatment with pembrolizumab.( The setting of 16 times administration is the period of adjuvant therapy of this trial is 12 month(=48weeks), administration of pembrolizumab is Q3W, so 16 times administration comes to 48 weeks.)
  Other Names: MK-3475; Keytruda

SUMMARY:
The aim of this study is to elucidate the utility of the immune checkpoint inhibitor pembrolizumab in preventing the recurrence of HCC when administered before and after curative surgery or ablation.

DETAILED DESCRIPTION:
Each subject will participate in the trial from the time he or she signs the informed consent form until the final contact. After a screening phase of up to 28 days, each subject will receive administration of pembrolizumab 200mg IV once only before curative treatment such as hepatic resection or radiofrequency ablation, and will receive curative treatment after administration of pembrolizumab. After curative treatment, each subject will receive pembrolizumab 200mg IV every 3 weeks. Treatment will continue until tumor recurrence, occurrence of an unacceptable adverse event, or the 16th treatment with pembrolizumab.( The setting of 16 times administration is the period of adjuvant therapy of this trial is 12 month(=48weeks), administration of pembrolizumab is Q3W, so 16 times administration comes to 48 weeks.) Subjects who discontinue for reasons other than tumor recurrence will have post-treatment follow-up visits for monitoring disease status until tumor recurrence, until initiation of non-study cancer treatment, until withdrawal of consent for study participation, or until becoming lost to follow-up. All subjects will be followed for overall survival until death, withdrawal of consent for study participation, or the end of the study, whichever comes first. After the end of trial treatment, each subject will be followed for 30 days for adverse event monitoring. Serious adverse events will be collected for 90 days after the end of treatment or for 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma for which radical cure is possible by resection or RFA.
* Diagnosed with typical HCC based on imaging findings with Intermediate or High Risk of recurrence as assessed by tumor characteristics.
* Male or female subjects >/= 20 years of age
* Child-Pugh score A
* ECOG Performance Status of 0.
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Recurrent HCC
* HCC with extrahepatic metastasis and/or vascular invasion confirmed by diagnostic imaging
* Subjects with poorly controlled ascites (excluding cases that responded to diuretic therapy)
* Subjects with hepatic encephalopathy
* Past history of immunotherapy
* Past history or complication of an active autoimmune disorder.
* Past history or complication of interstitial pneumonia.
* Past or current history of malignant tumor, except for curative cases
* Subjects with renal insufficiency requiring hemodialysis or peritoneal dialysis.
* Past or current history of severe cardiovascular disease
* Active clinically serious infections except for HBV or HCV
* Subjects with convulsive disorder requiring treatment (risk of convulsive seizures).
* Subjects with gastrointestinal bleeding causing clinical problems within a 4-week period before enrollment in this study.
* Subjects with thrombosis or embolism that developed within a 6-month period before enrollment in this study
* Subjects with pregnant or breast feeding, or planning to become a parent
* Subjects with possible allergic reaction to the investigational drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-10 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
One-year recurrence-free survival rate | 1 year after curative treatment
  One-year recurrence-free survival rate is defined as the recurrence-free survival rate 1year after curative treatment.

SECONDARY OUTCOMES:
Recurrence free survival | From the date of enrollment until the date of first recurrence or date of death from any cause, whichever came first, up to 72 weeks.
  Recurrence-free survival is defined as the length of time from the date of confirmation of complete cure to the earliest of the following: the date when recurrence is diagnosed or the date of death due to any cause.
Overall survival | From date of enrollment until the date of death from any cause, up to 72 weeks.
  Overall survival is defined as the length of time from the date of confirmation of complete cure to the date of death due to any cause.
Objective response rate after neoadjuvant phase | Evaluation period is just before curative treatment, up to 4 weeks.
  Tumor assessment in accordance with RECIST1.1 will be performed after neoadjuvant administration.
Tumor markers | From the date of enrollment until the date of last administration of study drug, up to 72 weeks.
  Baseline levels of tumor markers including AFP, AFP-L3, and PIVKA-II and changes in their levels will be exploratory investigated in relation to the therapy efficacy.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the date of enrollment until the date of last administration of study drug, thereafter up to 4 months
  The safety endpoints of this study are the safety of pembrolizumab as neoadjuvant and/or adjuvant therapy in patients with HCC. To determine the safety of the drug, the degree of toxicity is evaluated in accordance with the CTCAE (version 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Kudo, Professor, Principal Investigator — Kindai University Faculty of Medicine, Gastroenterology and Hepatology

IPD SHARING:
Plan to Share IPD: Undecided